CLINICAL TRIAL: NCT01083602
Title: A Phase II, Multi-center, Single Arm, Open Label Study of Panobinostat in Combination With Bortezomib and Dexamethasone in Patients With Relapsed and Bortezomib-refractory Multiple Myeloma
Brief Title: Efficacy of Panobinostat in Patients With Relapsed and Bortezomib-refractory Multiple Myeloma
Acronym: MACS1271
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589DUS71
Record Dates: First submitted 2010-03-08; First posted 2010-03-10 (Estimated); Results first posted 2015-03-27 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2017-11

CONDITIONS: Relapsed and Bortezomib Refractory Multiple Myeloma; Refractory Multiple Myeloma; Multiple Myeloma in Relapse
Keywords: Multiple Myeloma; Relapsed Multiple Myeloma; Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Panobinostat; Bortezomib; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- panobinostat + bortezomib & dexamethasone (Experimental): panobinostat in combination with bortezomib and dexamethasone in patients with relapsed and bortezomib-refractory multiple myeloma
  Interventions: Drug: panobinostat; Drug: bortezomib; Drug: dexamethasone

INTERVENTIONS:
Drug: panobinostat — PAN 20 mg PO given TIW, weeks 1&2 of each 3-week cycle;• BTZ 1.3 mg/m2 IV push given BIW weeks 1&2 of each 3 week cycle (days 1,4,8 and 11);• Dex 20 mg PO given QIW, weeks 1&2 of each 3-week cycle (days 1,2,4,5,8,9,11 and 12)
  Other Names: LBH589; PAN
Drug: bortezomib
  Other Names: BTZ
Drug: dexamethasone
  Other Names: DEX

SUMMARY:
This study is designed to assess the effectiveness of the combination of Panobinostat plus Bortezomib and Dexamethasone in patients with relapsed and bortezomib refractory Multiple Myeloma.

DETAILED DESCRIPTION:
This is a phase II, two stage, single arm, open label, multi-center study of oral PAN in combination with BTZ/Dex in patients with relapsed and refractory multiple myeloma, who are bortezomib-refractory and have received at least 2 prior lines of therapy. Patients must have been exposed to an iMID (lenalidomide or thalidomide) and progressed on or within 60 days of their last BTZ-containing line of therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a previous diagnosis of multiple myeloma, based on IMWG 2003 definitions. All three of the following criteria must have been met:

   * Monoclonal immunoglobulin (M component) on electrophoresis, and on immunofixation on serum or on total 24 hour urine
   * Bone marrow (clonal) plasma cells ≥ 10% or biopsy proven plasmacytoma
   * Related organ or tissue impairment (CRAB symptoms: anemia, hypercalcemia, lytic bone lesions, renal insufficiency, hyperviscosity, amyloidosis or recurrent infections)
2. Patient must have relapsed and refractory MM and must require treatment for the relapsed disease
3. Patients must have received at least 2 prior lines of therapy which include an IMiD (thalidomide or lenalidomide)
4. Patient must be refractory to the last bortezomib containing line of therapy given in the relapsed and refractory setting defined as:

   * having progressed on or within 60 days of the last bortezomib-containing line of therapy
5. Patient has measurable disease on M protein at study screening defined by at least one of the following measurements as per thresholds clarified in IMWG 2003 disease definitions (Kyle, et al 2003):

   * Serum M-protein ≥ 1 g/dL (≥ 10 g/L)
   * Urine M-protein ≥ 200 mg/24 h
6. Patients treated with local radiotherapy with or without concomitant exposure to steroids for pain control or management of cord/nerve root compression, are eligible. Two weeks must have lapsed since last date of radiotherapy, which is recommended to be a limited field. Patients who require concurrent radiotherapy should have entry to the protocol deferred until the radiotherapy is completed and 2 weeks have passed since the last date of therapy
7. Patient's age is ≥ 18 years at time of signing the informed consent
8. Patient has an Eastern Cooperative Oncology Group (ECOG) performance status (PS) of ≤ 2
9. Patient has the following laboratory values within 3 weeks before starting study drug (lab tests may be repeated, as clinically indicated, to obtain acceptable values before screen fail is concluded but supportive therapies are not to be administered within the week prior to screening tests for absolute neutrophil count or platelet counts)

   * Absolute neutrophil count (ANC) ≥ 1.0 x 109 /L
   * Platelet count ≥ 70 x 109 /L
   * Serum potassium, magnesium, phosphorus, within normal limits (WNL) for institution
   * Total calcium (corrected for serum albumin) or ionized calcium ≥ LLN, and not higher than CTCAE grade 1 in case of elevated value

   Note: Potassium, calcium, magnesium, and/or phosphorus supplements may be given to correct values that are < LLN:
   * AST/SGOT and ALT/SGPT ≤ 2.5 x ULN
   * Serum total bilirubin ≤ 1.5 ULN (or ≤ 3.0 x ULN if patient has Gilbert syndrome)
   * Serum creatinine levels ≤ 2.5 x ULN, or calculated creatinine clearance ≥ 40 ml/min
10. Patient has provided written informed consent prior to any screening procedures
11. Patient is able to swallow capsules
12. Patient must be able to adhere to the study visit schedule and other protocol requirements
13. Women of childbearing potential (WOCBP) must have a negative serum pregnancy test at within 7 days prior to start of study treatment

Exclusion Criteria:

1. Primary refractory disease (patients that never reached at least an MR for over 60 days under any prior therapy)
2. Patients who have a history of prior MM treatment with a DAC inhibitor including panobinostat
3. Patients who have had prior allogeneic stem cell transplantation and show evidence of active graft-versus-host disease that requires immunosuppressive therapy
4. Peripheral neuropathy ≥ CTCAE grade 2
5. Patients who will need valproic acid for any medical condition during the study or within 5 days prior to the first administration of study drug / treatment or who cannot be switch to safely to alternative anti-epileptic medication
6. Patients who have impaired cardiac function including any of the following:

   * Congenital long QT syndrome, complete left bundle branch block or use of a permanent cardiac pacemaker, history or presence of ventricular tachyarrhythmias, clinically significant resting bradycardia (< 50 beats per minute). Right bundle branch block + left anterior hemiblock (bifascicular block)
   * QTcF > 450 msec on screening ECG
   * Presence of unstable atrial fibrillation. Patients with stable atrial fibrillation are allowed in the study provided they do not meet other cardiac or prohibited drug exclusion criteria
   * Previous history of angina pectoris or acute MI within 6 months
   * Congestive heart failure (New York Heart Association functional classification III-IV)
   * Patient has any other clinically significant cardiovascular disease (e.g. uncontrolled hypertension)
7. Patient has an impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of panobinostat (e.g., ulcerative disease, uncontrolled nausea, vomiting, malabsorption syndrome, obstruction, or significant small bowel resection)
8. Patient has unresolved diarrhea ≥ CTCAE grade 2
9. Patients who have any other concurrent severe and/or uncontrolled medical condition(s) including, but not limited to: uncontrolled diabetes mellitus, active or uncontrolled infection, chronic obstructive or chronic restrictive pulmonary disease (e.g. dyspnea at rest from any cause), symptomatic thyroid dysfunction, significant bleeding tendency, that could cause unacceptable safety risks or compromise compliance with the protocol
10. Patients who are using medications that have a known relative risk of prolonging the QT interval or of inducing Torsade de Pointes, where such treatment cannot be discontinued or switched to a different medication prior to starting study drug
11. Women who are pregnant or breast feeding
12. Patients with evidence of another malignancy not in remission or history of such a malignancy within the last 5 years (except for treated basal or squamous cell carcinoma, or in situ cancer of the cervix)
13. Patients who have received prior to starting study treatment either radiation therapy to > 30% of marrow-bearing bone within 4 weeks; myelotoxic chemotherapy within 4 weeks; or immunotherapy within 8 weeks; or who have not yet recovered from side effects of such therapies
14. Patients with any significant history of non-compliance to medical regimens or unwilling or unable to comply with the instructions given to him/her by the study staff
15. Use of chemo-, biologic or immunologic therapy and/or other investigational agents while the patient is on study treatment.
16. Patient taking any anti-cancer therapy concomitantly (bisphosphonates are permitted only if commenced prior to the start of screening period)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2010-06; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals; Steven Young, M.D., Principal Investigator — Somerset Hematology Oncology
Locations (13):
- United States (13):
  - University of California at Los Angeles, Los Angeles, California
  - Stanford University Medical Center Division of Hematology, Stanford, California
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University School of Medicine/Winship Cancer Institute Dept. of Winship Cancer Inst., Atlanta, Georgia
  - Georgia Regents University MedCollege of GA Cancer Ctr 2, Augusta, Georgia
  - Hematology/Oncology of the North Shore Orchard Healthcare Res. Inc., Skokie, Illinois
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Somerset Hematology Oncology Associates Somerset Hema Oncol Assoc (2), Somerset, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Duke University Medical Center Dept. of DUMC (4), Durham, North Carolina
  - Vanderbilt University Medical Center, Clinical Trials Center Vanderbilt UMC, Nashville, Tennessee
  - MD Anderson Cancer Center/University of Texas MD Anderson CC, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Richardson PG, Schlossman RL, Alsina M, Weber DM, Coutre SE, Gasparetto C, Mukhopadhyay S, Ondovik MS, Khan M, Paley CS, Lonial S. PANORAMA 2: panobinostat in combination with bortezomib and dexamethasone in patients with relapsed and bortezomib-refractory myeloma. Blood. 2013 Oct 3;122(14):2331-7. doi: 10.1182/blood-2013-01-481325. Epub 2013 Aug 15. PMID 23950178

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Panobinostat + Bortezomib & Dexamethasone
Started | 55
Completed | 0
Not Completed | 55
Not completed — Adverse Event | 11
Not completed — New Cancer Therapy | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 5
Not completed — Lack of Efficacy | 36

BASELINE CHARACTERISTICS:
Population: The study population consisted of adult patients with relapsed and bortezomib-refractory MM who had received at least 2 prior lines of therapy and had been exposed to an IMiD (thalidomide or lenalidomide). Bortezomib-refractory was defined as demonstrated disease progression on or within 60 days of the last bortezomib -containing line of therapy.
Arm/Group | Panobinostat + Bortezomib & Dexamethasone
Number analyzed (Participants) | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (10.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 29

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (PR+nCR+CR)
Description: Overall response rate=(PR+nCR+CR) CR= < 5% plasma cells in bone marrow. No confirmation on bone marrow plasma cell (additional assessment) is needed to document CR except patients with non-secretory myeloma where the bone marrow examination must be repeated after an interval of at least 6 weeks, Absence of M-protein in serum and urine by immunofixation,nCR same as CR without out Absence of M-protein in serum and urine by immunofixation,PR+ 50% reduction of serum M-protein and sofft tissue Plasmacytomas all for more than 6 weeks.
Time Frame: after eight cycyles of treatment (24 weeks)
Population: Full Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Panobinostat + Bortezomib & Dexamethasone
Number analyzed (Participants) | 55
percentage of participants | 34.5 [22.2 to 46.7]

2. Secondary Outcome: Responders to Treatment
Description: The primary endpoint for this phase II study of patients with bortezomib-refractory MM is response after a maximum of 8 cycles of therapy as defined by the modified EBMT criteria.
Time Frame: after eight cycyles of treatment (24 weeks)
Population: Full Analysis Set
Measure: Number; unit: participants
Arm/Group | Panobinostat + Bortezomib & Dexamethasone
Number analyzed (Participants) | 55
participants
  Complete Response (CR) | 0 [22.2 to 46.7]
  near Complete Response(nCR) | 1
  Partial Response (PR) | 18
  Minimal Response (MR) | 10
  No Change | 20
  Pregressive Disease (PD) | 3
  Unknown | 3

3. Secondary Outcome: Time to Response (Greater Than or Equal to PR) Based on Investigator Assessment
Description: Time to response is defined as the time from the date of first administration of study treatment to the date of first documented evidence of CR or nCR or PR (whichever status is recorded first). Patients who do not have a response of PR or better by the data cut-off date are censored.
Time Frame: after eight cycyles of treatment (24 weeks)
Population: FAS
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Panobinostat + Bortezomib & Dexamethasone
Number analyzed (Participants) | 55
Days | 51.8 (30.92)

4. Secondary Outcome: Progression-free Survival
Description: Progression-free survival (PFS) was defined as the time from the date of first study treatment to first occurrence of documented progressive disease /relapse or death. Time from randomization until disease progression or death by Kaplan-Meier estimates
Time Frame: 24 weeks
Population: Full Analysis Set (FAS)
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Panobinostat + Bortezomib & Dexamethasone
Number analyzed (Participants) | 55
days | 164.0 [107.0 to 204.0]

5. Secondary Outcome: Time to Progression
Description: Time from randomization until objective tumor progression; does not include deaths-- Kaplan-Meier estimates
Time Frame: 24 weeks
Population: FAS
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Panobinostat + Bortezomib & Dexamethasone
Number analyzed (Participants) | 55
Days | 164.0 [107.0 to 204.0]

6. Secondary Outcome: Over All Survival
Description: Kaplan Meier estimates- median time to event
Time Frame: 24 weeks
Population: FAS
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Panobinostat + Bortezomib & Dexamethasone
Number analyzed (Participants) | 55
Days | 559.0 [329.0 to 682.0]

ADVERSE EVENTS:
Groups:
- PAN + BTZ + Dex: PAN + BTZ + Dex
Arm/Group | PAN + BTZ + Dex
Serious Adverse Events (participants affected / at risk) | 39/55
Other Adverse Events (participants affected / at risk) | 53/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PAN + BTZ + Dex (N=55)
Anaemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Pancytopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Atrial fibrillation (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 3
Diverticulum (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 2
Pyrexia (General disorders) | 5
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Hepatic ischaemia (Hepatobiliary disorders) | 1
Arthritis bacterial (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Clostridium difficile infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 2
Parainfluenzae virus infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 8
Postoperative wound infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 4
Septic shock (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Staphylococcal sepsis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 1
White blood cell count decreased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Hypophagia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Lethargy (Nervous system disorders) | 1
Peroneal nerve palsy (Nervous system disorders) | 1
Alcoholism (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 4
Renal impairment (Renal and urinary disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 3
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PAN + BTZ + Dex (N=55)
Anaemia (Blood and lymphatic system disorders) | 23
Neutropenia (Blood and lymphatic system disorders) | 11
Thrombocytopenia (Blood and lymphatic system disorders) | 23
Lacrimation increased (Eye disorders) | 5
Vision blurred (Eye disorders) | 10
Abdominal discomfort (Gastrointestinal disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 8
Abdominal pain upper (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 19
Diarrhoea (Gastrointestinal disorders) | 39
Dyspepsia (Gastrointestinal disorders) | 6
Flatulence (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 33
Stomatitis (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 16
Asthenia (General disorders) | 10
Chest pain (General disorders) | 3
Chills (General disorders) | 4
Fatigue (General disorders) | 37
Oedema (General disorders) | 6
Oedema peripheral (General disorders) | 21
Pyrexia (General disorders) | 8
Candida infection (Infections and infestations) | 3
Oral candidiasis (Infections and infestations) | 3
Rhinitis (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Tooth infection (Infections and infestations) | 3
Upper respiratory tract infection (Infections and infestations) | 18
Urinary tract infection (Infections and infestations) | 4
Contusion (Injury, poisoning and procedural complications) | 6
Fall (Injury, poisoning and procedural complications) | 3
Blood creatinine increased (Investigations) | 6
Weight decreased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 23
Dehydration (Metabolism and nutrition disorders) | 6
Hyperglycaemia (Metabolism and nutrition disorders) | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 13
Hypomagnesaemia (Metabolism and nutrition disorders) | 7
Hyponatraemia (Metabolism and nutrition disorders) | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 4
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 9
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 9
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Amnesia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 21
Dysgeusia (Nervous system disorders) | 13
Headache (Nervous system disorders) | 12
Hypoaesthesia (Nervous system disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 15
Paraesthesia (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 3
Syncope (Nervous system disorders) | 5
Tremor (Nervous system disorders) | 4
Confusional state (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 19
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Dry skin (Skin and subcutaneous tissue disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 8
Rash (Skin and subcutaneous tissue disorders) | 4
Skin lesion (Skin and subcutaneous tissue disorders) | 3
Deep vein thrombosis (Vascular disorders) | 4
Haematoma (Vascular disorders) | 3
Hot flush (Vascular disorders) | 4
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 9
Orthostatic hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.